CLINICAL TRIAL: NCT01439204
Title: A Randomized, Open-label, Parallel-Group, Single-dose, Biocomparability Study of the Pharmacokinetics of Abatacept (BMS-188667) Drug Products Using Active Pharmaceutical Ingredient Manufactured at Devens, MA Site Relative to Active Pharmaceutical Ingredient Manufactured at Lonza, New Hampshire (NH) in Healthy Subjects
Brief Title: Pharmacokinetic Study to Compare the Blood Levels of Abatacept Manufactured at Lonza Biologics to the Blood Levels of Abatacept Manufactured at the Devens, Massachusetts (MA) Facility of Bristol-Myers Squibb
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IM101-292
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abatacept (BMS-188667) manufactured at Lonza, NH facility (Active Comparator)
  Interventions: Biological: Abatacept (BMS-188667)
- Abatacept (BMS-188667) manufactured at Devens, MA facility (Experimental)
  Interventions: Biological: Abatacept (BMS-188667)

INTERVENTIONS:
Biological: Abatacept (BMS-188667) — Solution for injection, Intravenous, 750 mg, Single dose, 1 day,
  Other Names: BMS-188667

SUMMARY:
The purpose of this study is to determine whether the blood levels of Abatacept (BMS-188667) drug product manufactured at Lonza Biologics and the Devens, MA facility of Bristol-Myers Squibb are comparable in healthy subjects

DETAILED DESCRIPTION:
Primary Purpose of this study is to compare the pharmacokinetic (PK) of Abatacept (BMS-188667) manufactured at Lonza relative to Abatacept (BMS-188667) manufactured at Devens, MA facility following a single intravenous infusion of 750 mg in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, electrocardiograms (ECGs), and clinical laboratory determinations
* Body weight will be between 60 and 100 kg, inclusive

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Any major surgery within 4 weeks of study drug administration
* Smoking more than 10 cigarettes per day
* Recent (within 6 months of study drug administration) drug or alcohol abuse.
* Positive blood screen for hepatitis C antibody, hepatitis B surface antigen, or Human Immunodeficiency Virus-1, Human Immunodeficiency Virus-2 antibody
* History of any significant drug allergy or asthma
* Women who are pregnant or breastfeeding and/or unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 223 (Actual)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Icon Clinical Pharmacology Unit, Llc, Omaha, Nebraska, United States

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 October 2011 to 11 Feb 2012. Participants who were randomized to an arm were admitted to a clinical facility the day prior to dosing (Day -1) and confined until 24 hours post the single dose; participants followed to Day 71.
Pre-assignment Details: Healthy participants who weighed between 60 and 100 kilograms, inclusive. 223 enrolled; 72 randomized to an arm. Reasons for not being randomized: 24 withdrew consent, 5 poor/non-compliance, 111 no longer met study criteria, 11 other. Participants were age and sex matched between treatment arms.
Groups:
- 750 mg Abatacept From Lonza, NH: A single dose of abatacept 750 mg, manufactured at Lonza, New Hampshire facility, was administered intravenously (IV) using a calibrated, constant rate infusion pump over approximately 30 minutes.
- 750 mg Abatacept From Devens, MA: A single dose of abatacept 750 mg, manufactured at Devens, Massachusetts facility, was administered intravenously (IV) using a calibrated, constant rate infusion pump over approximately 30 minutes.
Period: Overall Study
Arm/Group | 750 mg Abatacept From Lonza, NH | 750 mg Abatacept From Devens, MA
Started | 36 | 36
Completed | 32 | 33
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — No longer meets study criteria | 1 | 0
Not completed — poor/non-compliance | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 750 mg Abatacept From Lonza, NH | 750 mg Abatacept From Devens, MA | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (10.02) | 31.2 (8.90) | 31.4 (9.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 14 | 15 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 32 | 30 | 62
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 36 | 36 | 72
Body Weight [Mean (Standard Deviation); unit: kg] — An inclusion criterion was that participants would weigh between 60 and 100 kilograms (kg), inclusive.
  kg | 78.93 (11.472) | 79.39 (11.057) | 79.16 (11.189)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of Single Dose Abatacept - Pharmacokinetic Evaluable Population
Description: Cmax was derived from serum concentration versus time data. Serum samples were analyzed for abatacept by a validated enzyme-linked immunosorbent assay (ELISA) and were obtained at: predose (0 hours), 0.25 hours (h), 0.5, 1, 2, 6, 12, 24, 72, 168, 336, 504, 672, 1008, 1344, and 1688 h post dose (Days 1 to 71). The results were summarized. The lower limit of assay quantitation (LLOQ) was 1.00 nanograms per milliliter (ng/mL). Cmax was measured in micro grams per milliliter (µg/mL).
Time Frame: Days 1 to 71
Population: Pharmacokinetic (PK) population: all participants who received study drug and had adequate PK profiles. All completers had evaluable PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | 750 mg Abatacept From Lonza, NH | 750 mg Abatacept From Devens, MA
Number analyzed (Participants) | 32 | 33
µg/mL | 262 (27) | 255 (21)

2. Primary Outcome: Time to Reach Maximum Concentration (Tmax) of Single Dose Abatacept - Pharmacokinetic Evaluable Population
Description: Tmax was derived from serum concentration versus time data. Serum samples were analyzed for abatacept by a validated enzyme-linked immunosorbent assay (ELISA) and were obtained at: predose (0 hours), 0.25 hours (h), 0.5, 1, 2, 6, 12, 24, 72, 168, 336, 504, 672, 1008, 1344, and 1688 h post dose (Days 1 to 71). The results were summarized. The lower limit of assay quantitation (LLOQ) was 1.00 nanograms per milliliter (ng/mL). Tmax was measured in hours (h).
Time Frame: Day 1 to Day 71
Population: Pharmacokinetic (PK) population: all participants who received study drug and had adequate PK profiles.
Measure: Median (Full Range); unit: h
Arm/Group | 750 mg Abatacept From Lonza, NH | 750 mg Abatacept From Devens, MA
Number analyzed (Participants) | 32 | 33
h | 1.00 [0.55 to 2.12] | 1.00 [1.00 to 6.00]

3. Primary Outcome: Area Under the Concentration-time Curve (AUC) From Time Zero to 28 Days [AUC(0-28 Days)] of Single Dose Abatacept - Pharmacokinetic Evaluable Population
Description: AUC (0 - 28) was derived from serum concentration versus time data. Serum samples were analyzed for abatacept by a validated enzyme-linked immunosorbent assay (ELISA) and were obtained at: predose (0 hours), 0.25 hours (h), 0.5, 1, 2, 6, 12, 24, 72, 168, 336, 504, 672, 1008, 1344, and 1688 h post dose (Days 1 to 71). The results were summarized. The lower limit of assay quantitation (LLOQ) was 1.00 nanograms per milliliter (ng/mL). AUC (0 - 28) was measured in micro grams*hours per milliliter (µg*h/mL).
Time Frame: Day 1 to Day 71
Population: Pharmacokinetic (PK) population: all participants who received study drug and had adequate PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | 750 mg Abatacept From Lonza, NH | 750 mg Abatacept From Devens, MA
Number analyzed (Participants) | 32 | 33
µg*h/mL | 33195 (26) | 35255 (23)

4. Primary Outcome: Area Under the Concentration-time Curve From Zero to the Last Time of the Last Quantifiable Concentration [AUC(0-T)] of Single Dose Abatacept - Pharmacokinetic Evaluable Population
Description: AUC (0 - T) was derived from serum concentration versus time data. Serum samples were analyzed for abatacept by a validated enzyme-linked immunosorbent assay (ELISA) and were obtained at: predose (0 hours), 0.25 hours (h), 0.5, 1, 2, 6, 12, 24, 72, 168, 336, 504, 672, 1008, 1344, and 1688 h post dose (Days 1 to 71). The results were summarized. The lower limit of assay quantitation (LLOQ) was 1.00 nanograms per milliliter (ng/mL). AUC (0 - T) was measured in micro grams*hour per milliliter (µg*h/mL).
Time Frame: Day 1 to Day 71
Population: Pharmacokinetic (PK) population: all participants who received study drug and had adequate PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | 750 mg Abatacept From Lonza, NH | 750 mg Abatacept From Devens, MA
Number analyzed (Participants) | 32 | 33
µg*h/mL | 39295 (23) | 41916 (25)

5. Primary Outcome: Area Under the Concentration-time Curve From Time Zero Extrapolated to Infinity [AUC(0 - INF)] of Single Dose Abatacept - Pharmacokinetic Evaluable Population
Description: AUC (0 - INF) was derived from serum concentration versus time data. Serum samples were analyzed for abatacept by a validated enzyme-linked immunosorbent assay (ELISA) and were obtained at: predose (0 hours), 0.25 hours (h), 0.5, 1, 2, 6, 12, 24, 72, 168, 336, 504, 672, 1008, 1344, and 1688 h post dose (Days 1 to 71). The results were summarized. The lower limit of assay quantitation (LLOQ) was 1.00 nanograms per milliliter (ng/mL). AUC (0 - INF) was measured in µg*h/mL.
Time Frame: Day 1 to Day 71
Population: Pharmacokinetic (PK) population: all participants who received study drug and had adequate PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | 750 mg Abatacept From Lonza, NH | 750 mg Abatacept From Devens, MA
Number analyzed (Participants) | 32 | 33
µg*h/mL | 40385 (23) | 43229 (27)

6. Primary Outcome: Terminal Phase Elimination Half-life (T-HALF) of Single Dose Abatacept - Pharmacokinetic Evaluable Population
Description: T-HALF was derived from serum concentration versus time data. Serum samples were analyzed for abatacept by a validated enzyme-linked immunosorbent assay (ELISA) and were obtained at: predose (0 hours), 0.25 hours (h), 0.5, 1, 2, 6, 12, 24, 72, 168, 336, 504, 672, 1008, 1344, and 1688 h post dose (Days 1 to 71). The results were summarized. The lower limit of assay quantitation (LLOQ) was 1.00 nanograms per milliliter (ng/mL). T-HALF was measured in hours (h).
Time Frame: Day 1 to Day 71
Population: Pharmacokinetic (PK) population: all participants who received study drug and had adequate PK profiles.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 750 mg Abatacept From Lonza, NH | 750 mg Abatacept From Devens, MA
Number analyzed (Participants) | 32 | 33
h | 344 (87.6) | 364 (106)

7. Primary Outcome: Total Body Clearance (CLT) of Single Dose Abatacept - Pharmacokinetic Evaluable Population
Description: CLT was the volume of abatacept cleared by the system, normalized by baseline body weight. Serum samples were analyzed for abatacept by a validated enzyme-linked immunosorbent assay (ELISA) and were obtained at: predose (0 hours), 0.25 hours (h), 0.5, 1, 2, 6, 12, 24, 72, 168, 336, 504, 672, 1008, 1344, and 1688 h post dose (Days 1 to 71). The results were summarized. The lower limit of assay quantitation (LLOQ) was 1.00 nanograms per milliliter (ng/mL). CLT was measured in milliliters per hours per kilogram of body weight (mL/h/kg).
Time Frame: Day 1 to Day 71
Population: Pharmacokinetic (PK) population: all participants who received study drug and had adequate PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h/kg
Arm/Group | 750 mg Abatacept From Lonza, NH | 750 mg Abatacept From Devens, MA
Number analyzed (Participants) | 32 | 33
mL/h/kg | 0.237 (24) | 0.219 (24)

8. Primary Outcome: Volume of Distribution at Steady-state (Vss) of Single Dose Abatacept - Pharmacokinetic Evaluable Population
Description: Vss was derived from serum concentration versus time data. Serum samples were analyzed for abatacept by a validated enzyme-linked immunosorbent assay (ELISA) and were obtained at: predose (0 hours), 0.25 hours (h), 0.5, 1, 2, 6, 12, 24, 72, 168, 336, 504, 672, 1008, 1344, and 1688 h post dose (Days 1 to 71). The results were summarized. The lower limit of assay quantitation (LLOQ) was 1.00 nanograms per milliliter (ng/mL). Vss was measured in liters per kg body weight (L/kg).
Time Frame: Day 1 to Day 71
Population: Pharmacokinetic (PK) population: all participants who received study drug and had adequate PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/kg
Arm/Group | 750 mg Abatacept From Lonza, NH | 750 mg Abatacept From Devens, MA
Number analyzed (Participants) | 32 | 33
L/kg | 0.088 (33) | 0.083 (22)

9. Secondary Outcome: Number of Participants With Positive Abatacept-induced Immunogenicity Response
Description: Immunogenicity determination was based on titers of anti-abatacept and anti- cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4-T) antibodies in serum over time. A participant had a positive abatacept-induced immunogenicity if 1 of the following criteria were met: missing baseline measurement and a positive response after baseline; negative baseline response and positive response after baseline; a baseline response and a positive response after baseline that has a titer value strictly greater than the baseline titer value. A validated, sensitive, electrochemiluminescence assay (ECL) method was used to analyze the antibodies in serum. Samples confirmed positive with ECL and with abatacept serum concentrations of less than equal to 1 µg/mL were further analyzed with a validated, in vitro, cell-based bioassay to analyze the sera containing the abatacept neutralizing activity. Samples obtained on Days 29, 57 and 71 post dose of abatacept on Day 1 (baseline).
Time Frame: Days 29, 57, 71
Population: Immunogenicity Data Set: All participants with at least 1 postdose visit.
Measure: Number; unit: participants
Arm/Group | 750 mg Abatacept From Lonza, NH | 750 mg Abatacept From Devens, MA
Number analyzed (Participants) | 36 | 36
participants | 4 | 1

10. Secondary Outcome: Number of Participants With Marked Serum Chemistry Abnormalities on Days 2, 15, 29, 57 and 71 - Safety Population
Description: Blood samples obtained: Days 1, 2, 4, 8, 15, 22, 29, 43, 57 and 71. International Units per liter (U/L); milligram per deciliter (mg/dL); Male(M); Female (F). Reference ranges (low/high) for laboratories for which participants were identified with marked abnormalities during the study: Blood Urea Nitrogen (M/F) 10-20mg/dL ; Creatine Kinase (F) 21-21 U/L,(M) 32-294 U/L; Direct Bilirubin (M/F) 0.1-0.4 mg/dL ; Fasting Glucose (M/F) 70-110 mg/dL; Lactate Dehydrogenase (M/F) 110-209 U/L.
Time Frame: Day 2 to Day 71
Population: All participants who received study drug (safety population) and had a laboratory assessment were included in the analysis. Day 2 N=36 both arms; Day 15 (Lonza arm N=36; Devens arm N=34; Day 29 (Lonza arm N=34; Devens arm N=33); Day 57 (Lonza arm N=31; Devens arm N=33); Day 71 (Lonza arm N=36; Devens arm N=34).
Measure: Number; unit: participants
Arm/Group | 750 mg Abatacept From Lonza, NH | 750 mg Abatacept From Devens, MA
Number analyzed (Participants) | 36 | 36
participants
  Creatine Kinase (high) Day 2 (N=36) | 1 | 0
  Creatine Kinase (high) Day 15 (N=36,34) | 1 | 0
  Creatine Kinase (high) Day 29 (N=34,33) | 2 | 1
  Creatine Kinase (high) Day 57 (N=31,33) | 1 | 1
  Creatine Kinase (high) Day 71 (N=36,34) | 1 | 2
  Lactate Dehydrogenase (high) Day 2 (N=36) | 0 | 1
  Blood urea nitrogen (high) Day 15 (N=36,34) | 1 | 0
  Blood urea nitrogen (high) Day 29 (N=34) | 0 | 1
  Blood urea nitrogen (high) Day 71 (N=36,34) | 2 | 0
  Bilirubin Direct (high) Day 29 (N=34) | 0 | 3
  Bilirubin Direct (high) Day 71 (N=36,34) | 0 | 1
  Fasting Glucose (high) Day 71 (N=36,34) | 1 | 0

11. Secondary Outcome: Number of Participants With Marked Hematology Abnormalities on Days 2, 15, 29, 57, and 71 - Safety Population
Description: Blood samples obtained: Days 2, 4, 8, 15, 22, 29, 43, 57 and 71. Male(M); Female (F). Reference ranges (low/high) for laboratory parameters for which participants were identified with marked abnormalities during the study: Leukocytes (quantitative White blood cells) (M/F) 4-11*10^3/microliters (µL); Neutrophils (absolute)(M/F) 1.4- 8.2*10^3/µL.
Time Frame: Day 2 to Day 72
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | 750 mg Abatacept From Lonza, NH | 750 mg Abatacept From Devens, MA
Number analyzed (Participants) | 36 | 36
participants
  Any marked abnormalities Day 2 (N=36) | 0 | 0
  Any marked abnormalities Day 15 (n=36,34) | 0 | 0
  Leukocytes (high) Day 29 (N=34,33) | 0 | 1
  Leukocytes (high) Day 57 (N=31,33) | 0 | 1
  Leukocytes (high) Day 71 (N=36,34) | 1 | 1
  Neutrophils (absolute) (high) Day 71 (N=36,34) | 1 | 1

12. Secondary Outcome: Change From Baseline in Systolic Blood Pressure - Safety Population
Description: Blood pressure was obtained while the participant had been quietly seated for at least 5 minutes. Baseline was the 0 hour measurement on Day 1 (day of dosing) or if this value was missing, the last measurement before dosing. Blood pressure was measured in millimeters of mercury (mmHg) on Days 1, 2, 15, 29, 57, and 71.
Time Frame: Day 1 to Day 71
Population: All participants who received study drug (safety population) and had systolic assessment were included in the analysis. Days 1 and 2 N=36 both arms; Day 15 (Lonza arm N=36; Devens arm N=34; Day 29 (N=33 in both arms); Day 57 (Lonza arm N=31; Devens arm N=33); Day 71 (Lonza arm N=36; Devens arm N=34).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 750 mg Abatacept From Lonza, NH | 750 mg Abatacept From Devens, MA
Number analyzed (Participants) | 36 | 36
mmHg
  Day 1 (1 hour post dose) (N=36) | -6.3 (9.73) | -4.5 (9.06)
  Day 2 (N=36) | -3.0 (12.31) | -1.4 (10.35)
  Day 15 (N=36,34) | -1.1 (12.09) | 0.3 (8.12)
  Day 29 (N=33) | -2.3 (10.94) | -0.2 (9.65)
  Day 57 (N=31,33) | 1.0 (11.96) | 3.4 (9.48)
  Day 71 (N=36,34) | 2.2 (12.09) | 2.9 (9.87)

13. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure on Days 1, 2, 15, 29, 57, and 71 - Safety Population
Description: as for outcome 12
Time Frame: Day 1 to Day 71
Population: All participants who received study drug (safety population) and had diastolic assessment were included in the analysis. Day 2 N=36 both arms; Day 15 (Lonza arm N=36; Devens arm N=34; Day 29 (N=33 in both arms); Day 57 (Lonza arm N=31; Devens arm N=33); Day 71 (Lonza arm N=36; Devens arm N=34).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 750 mg Abatacept From Lonza, NH | 750 mg Abatacept From Devens, MA
Number analyzed (Participants) | 36 | 36
mmHg
  Day 1 (1 hour post dose) N=36 | -4.9 (5.91) | -4.1 (5.78)
  Day 2 (N=36) | -2.3 (8.98) | -0.6 (6.02)
  Day 15 (N=36,34) | -1.4 (7.45) | 1.0 (7.29)
  Day 29 (N=33) | -1.9 (6.37) | 0.9 (7.08)
  Day 57 (N=31,33) | 0.4 (7.48) | 3.5 (7.56)
  Day 71 (N=36,34) | 1.6 (8.59) | 4.0 (5.78)

14. Secondary Outcome: Number of Participants With a Change From Baseline in QT Interval and Corrected (Fridericia) QT Interval (QTcF) - Safety Population
Description: 12-lead electrocardiograms were performed on a supine participant (5 minutes supine) at baseline (baseline = screening; Days -21 to -2) and at Day 71. QT interval and QTc were measured in mille seconds (msec). A change from baseline QT and QTc (corrected for heart rate by Fridericia formula) greater than (>) 30 msec or less than (<) 60 msec were presented, as well as values over 450 and 500 msec. QT interval on ECG image defined as: time from the beginning of the QRS (complex consisting of Q, R and S waves) to the end of the T wave.
Time Frame: Day 1 to Day 71
Population: All participants who received study drug and had at least one ECG value.
Measure: Number; unit: participants
Arm/Group | 750 mg Abatacept From Lonza, NH | 750 mg Abatacept From Devens, MA
Number analyzed (Participants) | 36 | 36
participants
  Change from baseline in QT >60 msec | 0 | 1
  Change from baseline in QT >30 msec < 60 msec | 5 | 4
  Change from baseline in QTc >60 msec | 0 | 0
  Change from baseline in QTc >30 msec < 60 msec | 2 | 2
  QT > 500 msec | 0 | 0
  QT > 450 msec | 0 | 1
  QTcF >450 msec | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 71
Arm/Group | 750 mg Abatacept From Devens, MA | 750 mg Abatacept From Lonza, NH
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 11/36 | 12/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 750 mg Abatacept From Devens, MA (N=36) | 750 mg Abatacept From Lonza, NH (N=36)
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dizziness (Nervous system disorders) | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Vision blurred (Eye disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Headache (Nervous system disorders) | 5 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dysuria (Renal and urinary disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.